CLINICAL TRIAL: NCT06581393
Title: First Evaluation of the Moda-Flx Hemodialysis System™ in Real World Clinical Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diality Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIA-NSR-001
Record Dates: First submitted 2024-08-26; First posted 2024-09-03 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2024-08

CONDITIONS: End Stage Renal Disease; End Stage Renal Disease on Dialysis; End Stage Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Professional Care in an In-Center Hemodialysis Setting (Experimental): Hemodialysis using the Moda-flx Hemodialysis System
  Interventions: Device: Moda-flx Hemodialysis System

INTERVENTIONS:
Device: Moda-flx Hemodialysis System — All participants will complete up to 4 dialysis treatments on the Moda-flx Hemodialysis System over a period of up to 2 weeks.

SUMMARY:
This is a non-significant risk study utilizing a device cleared for use by the FDA under its 510(k) clearance. Consented patients will complete their usual dialysis treatment under professional care in an ICHD (In-Center Hemodialysis) setting.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of end stage kidney disease (ESKD) adequately treated by maintenance dialysis (defined as achieving a spKt/V ≥ 1.2 OR stdKt/V ≥ 2.1) and be deemed stable by their treating nephrologist prior to consent.
* Must sign the informed consent and a Health Insurance Portability and Accountability Act of 1996 (HIPAA) compliant authorization statement.
* Understand the nature of the procedures and the requirements of the Study.

Exclusion Criteria:

* Have a significant cognitive impairment that would preclude informed consent or the capacity for completing dialysis as prescribed by their treating nephrologist.
* In the opinion of the treating nephrologist, any other reason in which study participation would result in undue risk, including but not limited to protocol required prescription parameters.
* Are contraindicated for or not indicated to use the Moda-flx Hemodialysis System™ according to the Instructions For Use (IFU).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Single-Pool Standardized Dialysis Adequacy | Samples will be collected before and after each dialysis treatment at Visit 1, Visit 2, Visit 3 and at Visit 4 over a two week period
  Single-pool standardized dialysis adequacy (spKt/V) will be measured using the second-generation formula of Daugirdas. This formula normalizes urea clearance among heterogeneous hemodialysis schedules, where K=dialyzer clearance or urea, t=treatment time, and V=subject's volume of urea distribution. spKt/V values of ≥ 1.2 are regarded as being adequate.
Changes in Blood Chemistry | Samples will be collected at Visit 1 prior to initiating the first dialysis treatment, Visit 2, Visit 3 and at the conclusion of Visit 4 over a two week period
  Changes in overall blood chemistry laboratory levels from Visit 1 to Visit 4.
Changes in Complete Blood Count | Samples will be collected at Visit 1 prior to initiating the first dialysis treatment, Visit 2, Visit 3 and at the conclusion of Visit 4 over a two week period
  Changes in overall complete blood count levels from Visit 1 to Visit 4.
Changes in Iron Studies | Samples will be collected at Visit 1 prior to initiating the first dialysis treatment, Visit 2, Visit 3 and at the conclusion of Visit 4 over a two week period
  Changes in overall iron studies levels from Visit 1 to Visit 4.

CONTACTS AND LOCATIONS:
Locations (1):
- North America Research Institute, Ontario, California, United States

IPD SHARING:
Plan to Share IPD: No